CLINICAL TRIAL: NCT00006158
Title: AIDS Wasting in Women: Anabolic Effects of Testosterone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: anabole (completed); DK54167
Record Dates: First submitted 2000-08-08; First posted 2000-08-09 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: AIDS Wasting Syndrome
Keywords: AIDS; HIV; weight loss; Wasting Syndrome; testosterone; androgen levels; hormones
MeSH Terms: conditions — HIV Wasting Syndrome; Acquired Immunodeficiency Syndrome; Weight Loss; Wasting Syndrome | interventions — Testosterone

INTERVENTIONS:
Drug: Testosterone

SUMMARY:
The study is a 6 month, placebo-controlled study of transdermal testosterone for women with HIV-associated weight loss. Women with AIDS wasting have been found to have low testosterone levels. This study is designed to test the efficacy of physiologic testosterone dosing to improve weight, muscle mass and quality of life indices, including energy level, appetite and libido, in androgen deficient women with AIDS wasting. After 6 months, all women receive open label transdermal testosterone for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Females using acceptable form of birth control during study, including barrier contraception or IUD but excluding oral contraceptives or Depo-Provera
* Documented HIV infection
* Free testosterone level 3.0 pg/mL
* Weight < 90% or weight loss > 10% of pre-illness weight

Exclusion Criteria:

* Pregnant or actively seeking pregnancy
* Breast feeding
* New opportunistic infection diagnosed within 4 weeks of the study
* Requiring parenteral nutrition or pharmacologic glucocorticoid therapy
* Intractable diarrhea (6 stools/day)
* Androgen, estrogen, progestational derivative, or glucocorticoid administration within 3 months of the study, including Megace
* New retroviral therapy within 6 weeks of study
* SGOT > 5 X normal and/or clinically significant liver disease
* Creatinine > 2.0 mg/dL and/or clinically significant renal disease
* Hgb < 8.0 g/dL
* Active substance abuse or alcoholism

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1998-09; Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Miller K, Corcoran C, Armstrong C, Caramelli K, Anderson E, Cotton D, Basgoz N, Hirschhorn L, Tuomala R, Schoenfeld D, Daugherty C, Mazer N, Grinspoon S. Transdermal testosterone administration in women with acquired immunodeficiency syndrome wasting: a pilot study. J Clin Endocrinol Metab. 1998 Aug;83(8):2717-25. doi: 10.1210/jcem.83.8.5051. PMID 9709937
- [Background] Corcoran C, Grinspoon S. Treatments for wasting in patients with the acquired immunodeficiency syndrome. N Engl J Med. 1999 Jun 3;340(22):1740-50. doi: 10.1056/NEJM199906033402207. No abstract available. PMID 10352167